CLINICAL TRIAL: NCT00800774
Title: Ten-year Follow-up of Laser in Situ Keratomileusis in Patients 8 to 15 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARVO - BN - 2009
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2008-09

CONDITIONS: Anisometropia
Keywords: LASIK; safety; efficacy; stability; high anisometropia; patients 8 to 15 years old; conventional treatments have failed
MeSH Terms: conditions — Anisometropia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Nine eyes of nine patients (3 male and 6 female) with high anisometropia (>3.50 D), were included in this study. Minimum follow-up was 10 years. All patients were treated with the Chiron Technolas 217 excimer laser.
  Interventions: Procedure: LASIK

INTERVENTIONS:
Procedure: LASIK — Nine eyes of nine patients (3 male and 6 female) with high anisometropia (>3.50 D), were included in this study. Minimum follow-up was 10 years. All patients were treated with the Chiron Technolas 217 excimer laser.

SUMMARY:
The purpose of this study is to determine the safety, efficacy, predictability, and stability of laser in situ keratomileusis (LASIK) to correct high anisometropia in patients 8 to 15 years old in whom conventional treatments have failed.

DETAILED DESCRIPTION:
Nine eyes of nine patients (3 male and 6 female) with high anisometropia (>3.50 D), were included in this study. Minimum follow-up was 10 years. All patients were treated with the Chiron Technolas 217 excimer laser.

ELIGIBILITY:
Inclusion Criteria:

* High anisometropia (>3.50 D)
* Patients 8 to 15 years old
* Conventional treatments have failed

Exclusion Criteria:

* Diabetes
* Autoimmune diseases
* Topographic abnormalities

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 1998-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belquiz A Nassaralla, MD, PhD, Study Chair — Instituto de Olhos de Goiania
Locations (1):
- IOG, Goiânia, Goiás, Brazil